CLINICAL TRIAL: NCT02903771
Title: Phase I Study of Intra-peritoneal Cantrixil in Patients With Persistent or Recurrent Ovarian Cancer, Fallopian Tube Cancer or Primary Peritoneal Cancer.
Brief Title: Phase I Study of Cantrixil in Patients With Ovarian Cancer, Fallopian Tube Cancer or Primary Peritoneal Cancer.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kazia Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVGN-002-101
Record Dates: First submitted 2016-09-12; First posted 2016-09-16 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms
Keywords: Cantrixil; Intraperitoneal
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms | interventions — 4-(para-hydroxyphenyl)-7,4'-dihydroxy-3',5'-dimethoxy-8-methylisoflavan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Part A and Part B (Experimental): Part A (Dose Escalation):
  Part A is a Dose Escalation study to determine the Maximum Tolerated Dose of Cantrixil as a monotherapy.
  The tolerance of Cantrixil in combination with standard chemotherapy agents will also be examined.
  Part B (Expansion Cohort):
  An expansion cohort of an additional 12 patients will be recruited at the MTD.
  Interventions: Drug: Part A: Dose Escalation of Cantrixil; Drug: Part B: Expansion Cohort of Cantrixil

INTERVENTIONS:
Drug: Part A: Dose Escalation of Cantrixil — Cantrixil will be administered via the intraperitoneal route only. The dose of study drug that each participant will receive will depend on how far the study has progressed when the participant enrols. There are 9 potential doses of Cantrixil, they are 0.06, 0.12, 0.24 (starting dose), 0.6, 1.25, 2.5, 5, 10, or 20 mg/kg. The dose each participant receives will remain the same during the study, unless it needs to be reduced for safety reasons. The dose will not be increased.
  Each participant will receive the study drug once a week during the first two cycles; each cycle is 21-days (three weeks); the MTD will be determined during Cycle 1 only. If after two cycles of monotherapy, the patient tolerates Cantrixil adequately, they may continue to receive Cantrixil once a week and will also begin combination chemotherapy for another 6 cycles. Participants will receive no more than 8 cycles of study drug.
  Other Names: TRX-E-002-1 in 20% SBECD
Drug: Part B: Expansion Cohort of Cantrixil — Once the MTD has been established, an expansion cohort will be recruited at the MTD. An additional 12 patients will be recruited in this cohort on top of those recruited in Part A at the MTD. These patients will be subjected to the same intervention described in Part A with 2 cycles of monotherapy followed by up to 6 cycles of combination therapy.
  Other Names: TRX-E-002-1 in 20% SBECD

SUMMARY:
The main purpose of this study is to determine the safety and feasibility of weekly intra-peritoneal administration of Cantrixil to women with persistent or recurrent ovarian cancer, Fallopian tube cancer or primary peritoneal cancer. The study also aims to determine the maximum tolerated dose of Cantrixil in these patients when administered as a monotherapy or a combination therapy.

DETAILED DESCRIPTION:
This study is a progressive design with 2 discrete Parts (Part A: Dose escalation, Part B: Dose expansion. Cycle 1/Part A is a dose-finding assessment (dose escalation) to establish the maximum tolerated dose (MTD) of Cantrixil when administered as a single dose once a week for 3 weeks. Cycle2/Part A continues with 3 additional weekly doses of Cantrixil as a monotherapy before an assessment of disease response. In Cycles 3 to 8/Part A, patients will be administered the same once weekly dose of Cantrixil they tolerated in Cycles 1 and 2 (tolerance defined as no dose limiting toxicities [DLTs] or unacceptable treatment-related adverse events [AEs]) in combination with a limited range of standard chemotherapy agent(s), in order to assess the safety and tolerability of Cantrixil in combination therapy. Standard chemotherapy drugs will be administered at the standard efficacious doses to maintain optimum benefit of known drug combinations for patients.

Once the MTD has been determined in Part A, an additional 12 patients will be recruited in an expansion cohort for Part B. These patients will receive 2 cycles of Cantrixil monotherapy at the MTD, followed by up to 6 cycles of combination therapy.

Patients enrolled into the respective parts of the study may not receive treatments under different parts of the protocol.

To accommodate the intraperitoneal administration of Cantrixil, an in-dwelling, closed catheter or port will be inserted if the patient does not already have one. For intraperitoneal ports, the minimum period between port placement and the first administration of Cantrixil must not be shorter than 7 days.

Patients should begin protocol treatment within a maximum of 28 days of enrolment (i.e., signing of consent form).

Patients will start at Dose Level 0 which is calculated to be the human equivalent of 10% of the severely toxic dose in 10% (STD10) dose in rats (dose that is 1/10 the severely toxic dose in 10% of rats tested). Dose levels -1 and -2 will only be activated if there are 2 DLTs at the Dose Level 0 and -1, respectively. Single patient cohorts will be treated with increasing doses of Cantrixil until an AE is observed that meets the definition of a Dose Limiting Toxicity (DLT) or, in the opinion of the Data Safety Monitoring Committee (DSMC) and the Investigator, is causally related to study treatment and warrants observing additional patients at this dose level; at this point the study will revert to a 3+3 rules based dose escalation study. Once the study enters a 3+3 rules-based design, the study will not revert back to single patient cohorts.

If any unacceptable treatment-related AE or DLT is observed in any cycle, patients may be dose reduced to the next lower dose level of Cantrixil for subsequent doses of therapy. If a second unacceptable treatment-related AE or DLT is observed during any cycle within the same patient, treatment for the patient with Cantrixil will be discontinued. Investigators may continue with the standard chemotherapy at their discretion and if it is considered safe and in the patient's best interest.

If any of the following unacceptable treatment-related AEs or DLTs are observed and unless clearly unrelated to study treatment (e.g., disease progression), treatment at the allocated Cantrixil dose will be discontinued and dose escalation may be considered:

* Hematologic toxicity

  * Grade 4 neutropenia, lasting at least 5 days,
  * Grade 3 or Grade 4 neutropenia associated with fever >38.5°C,
  * Grade 4 thrombocytopenia lasting at least 5 days,
  * Grade 3 thrombocytopenia associated with severe bleeding in the opinion of the Investigator,
  * Dose delay of ≥3 weeks due to failure to recover counts.
* Any Common Terminology Criteria for Adverse Events (CTCCTCAE) version 4.03 Grade 3 or Grade 4 non haematological toxicity except:

  * Alopecia
  * Grade 3 abdominal pain deemed related to the port or catheter as determined by the treating physician
  * Grade 3 anorexia
  * Grade 3 fatigue
  * Grade 3 nausea and/or vomiting, or diarrhoea, lasting ≤48 hours with or without maximal medical management.
  * Grade 3 dehydration as a result of nausea and vomiting
  * Grade 3 constipation
  * Grade 3 metabolic abnormalities [hypokalaemia, hypomagnesemia, hypocalcaemia, hypophosphatemia]) that recovers to Grade 1 or less within 48 hours with or without medical management o• Other serious adverse events (SAEs) which, in the opinion of the treating Investigator, are related to investigational product and necessitate temporary or permanent cessation of administration o• Treatment delays of ≥3 weeks due to any treatment-related non-haematological toxicity will constitute a DLT All patients who discontinued from the study (i.e. are now Off Therapy/ End of Therapy) treatment will progress to follow-up unless the patient withdraws consent.

The initiation of each new cycle of Cantrixil will be at the discretion of the Investigator and will depend on the potential or measurable benefit to the patient assuming continued tolerability and adequate organ function.

Cantrixil treatment will be stopped due to RECIST version 1.1 defined disease progression observed after at least 4 cycles of therapy, recurrence of unacceptable toxicity after 1 Cantrixil dose reduction or patient consent withdrawal. Note that patients with progressive disease at the end of 2 cycles of Cantrixil monotherapy will not be taken off therapy if Cantrixil has been well tolerated. Pre-clinical data would suggest that the maximum benefit from Cantrixil will be realised as a combination therapy, hence all patients will have the opportunity to continue receiving Cantrixil as a combination therapy. Additionally, patients receiving combination therapy that are observed to have progressive disease as identified by RECIST version 1.1 criteria but who, in the opinion of the Investigator, continued to derive clinical benefit may continue Cantrixil treatment. Patients may also be discontinued from study treatment if the Investigator considers continuing therapy is not in the patient's best interest. All patients discontinued from study treatment will progress to follow-up unless the patient withdraws consent.

Tumour assessment via radiological imaging will be conducted during screening and every 6 weeks after the start of therapy, i.e. at the end of monotherapy and then after every 2 cycles of combination therapy. Either contrast-enhanced magnetic resonance imaging (MRI) or contrast-enhanced computed tomography (CT) may be used, but once a modality is used at baseline this must be used consistently for that patient throughout their participation on the study. Other imaging is not mandatory, but may be performed if clinically indicated.

Adverse events will be monitored for the duration of the study from the time of informed consent. Blood samples will be collected weekly for standard safety testing, or more frequently if clinically relevant, during the study. Additional volumes of blood will be collected before and after administration of Cantrixil for pharmacokinetic (PK) analysis (4 mL per time point as per the proposed PK schedule and for any exploratory studies (at baseline, end of Cycle 2 and end of treatment, 15 to 20 mL at each time-point).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have recurrent or persistent epithelial ovarian, fallopian tube, or primary peritoneal cancer. The original diagnosis must be verified by a histology report. All histological sub-types and all grades of disease are eligible to participate; grade, histological sub-type and breast cancer susceptibility gene (BRCA) status must be recorded at study entry.
2. Patients must be female and at least 18 years old.
3. Patients with malignant ascites are eligible to participate; paracentesis will be conducted before the administration of Cantrixil. Drainage of the maximum volume of ascites necessary for symptomatic relief should be performed according to local standard operating procedures before administration of Cantrixil.
4. Patients must have completed at least two (2) or more prior therapies (including adjuvant therapy) for their ovarian, Fallopian tube or primary peritoneal cancer prior to participation in the current study; all prior therapies must be recorded at baseline. Patients that have received prior intraperitoneal therapy are eligible for this study.
5. Patients must have platinum-resistant relapsed disease, platinum refractory disease, or have documented intolerance to platinum therapy. Patients will not be eligible based on rising CA-125 levels alone, patients must have other clinical symptoms (such as malignant ascites) or radiological tumour measurements that support disease recurrence or progression.
6. At least 4 weeks must have passed from any previous therapy and any toxicities from prior therapies (6 weeks for bevacizumab, nitrosoureas or mitomycin C treatment) must have resolved to less than or equal to Common Terminology Criteria for Adverse Events (CTCAE version 4.03) Grade 1 with the exception of alopecia, Grade 2 prior platinum-therapy related neuropathy and Grade 2 anaemia.
7. Patients must have a performance status of Eastern Cooperative Oncology Group (ECOG) 0 to 2 and, in the Investigator's opinion, be able to complete at least a major part of the study.
8. Patients must be willing and able to undergo insertion of a port or catheter for intraperitoneal access; the type of port or catheter used will be recorded.
9. Patients may have measurable or non-measurable disease; disease response and progression will be measured and assessed according to RECIST version 1.1 criteria using contrast CT, MRI and CA 125 measurements.
10. Patients must have acceptable hepatic and marrow function as defined below:

    * Absolute neutrophil count >1.5 x 109/L
    * Platelets >100 x 109/L
    * Total bilirubin; <2.5 times the institutional upper limit of normal (ULN)
    * Haemoglobin (Hb) of >10 g/dL; patients with Hb >9g/dL will be considered for this study if they have not received a transfusion or other bone marrow support. Patients with Hb >10 g/dL that have received a recent transfusion will only be eligible if there has been a wash-out period of 7 days for rhesus factor and 10 days for platelet transfusions, respectively.
    * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/ alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) ≤2.5 x institutional ULN.
    * Serum creatinine <1.5 x ULN
    * Prothrombin time (PT) or international normalised ratio (INR) ≤1.5 x ULN and activated partial thromboplastin time (aPTT) ≤1.5 x ULN if not on anticoagulation treatments.
11. Patients must be willing and able to comply with all study requirements, including treatment timing and/or nature of required assessments and treatment at designated study centre.
12. Each participant must be adequately informed about the purpose of the study; potential benefits and risks; their right to refuse participation or to withdraw consent at any time; institutional affiliation and potential competing interests of the researcher; and sources of study funding and have signed and dated a written informed consent form.

Exclusion Criteria:

1. Patients who have had chemotherapy, biologic therapy, immunotherapy, or radiotherapy within 4 weeks (6 weeks for bevacizumab, nitrosoureas or mitomycin C) prior to entering the study.
2. Patients must not have had major surgery within 4 weeks prior to screening.
3. Patients may not have received any other investigational medicinal products (IMPs) or participated in any other interventional clinical research studies within 3 months of the first Cantrixil administration.
4. Patients receiving any medications or substances that are strong inhibitors or inducers of cytochrome P450 (CYP)1A2, CYP2B6 and CYP3A4 or those substances with narrow therapeutic index are not to be enrolled. These compounds are prohibited from screening until completion of end of therapy or first post-treatment follow-up visit. For a list of prohibited medications see the University of Indiana Clinical Pharmacology Department's P450 Drug Interaction Table (http://medicine.iupui.edu/clinpharm/ddis/main-table/). Note: the use of paclitaxel is allowed, but only 24 hours after Cantrixil administration.
5. Patients at high risk of bowel perforation are excluded, including but not limited to any one or more of the following;

   * Patients with a recent history (previous 12 months) of bowel obstruction prior to study entry
   * Patients with CT scans that suggest invasion of bowel by tumour
   * Patients with symptoms to suggest impending bowel obstruction
   * Patients with prior whole abdominal radiotherapy
   * Patients with chronic inflammatory bowel diseases such as Crohn's disease or ulcerative colitis
6. Patients may not have uncontrolled or severe systemic diseases or psychiatric conditions, which in the treating physician's opinion makes it unsafe for the patient to participate in the study or would hinder compliance with the protocol. Screening for chronic conditions is not required.
7. Patients that are pregnant, lactating, or unable to adopt adequate contraception are excluded. Women of childbearing potential must have a negative pregnancy test within 7 days prior to screening.
8. Patients with a known history of hepatitis B or C.
9. Patients known to have tested positive for human immunodeficiency virus (HIV)
10. Patients with a known hypersensitivity to or serious reaction to benzopyrans are excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A/Prof Jermaine (Jim) Coward, MBBS FRACP PhD, Principal Investigator — ICON Cancer Care, Queensland, Australia; Dr Don Dizon, MD, FACP, Principal Investigator — Lifespan Cancer Institute, Rhode Island, USA
Locations (6):
- United States (3):
  - Peggy and Charles Stephenson Cancer Center, OU Health Sciences Center, Oklahoma City, Oklahoma
  - Lifespan Cancer Institute, Rhode Island Hospital, Providence, Rhode Island
  - Mary Crowley Cancer Research Center, Dallas, Texas
- Australia (3):
  - Westmead Adults Hospital, Westmead, New South Wales
  - ICON Cancer Care, South Brisbane, Queensland
  - Flinders Medical Centre, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Coward JI, Barve MA, Kichenadasse G, Moore KN, Harnett PR, Berg D, Garner JS, Dizon DS. Maximum Tolerated Dose and Anti-Tumor Activity of Intraperitoneal Cantrixil (TRX-E-002-1) in Patients with Persistent or Recurrent Ovarian Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer: Phase I Study Results. Cancers (Basel). 2021 Jun 26;13(13):3196. doi: 10.3390/cancers13133196. PMID 34206826

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 6 centres in 2 countries (USA and Australia) between December 2016 and March 2020. The first patient was enrolled on 05 December 2016 and the last patient was enrolled on 30 July 2019.
Pre-assignment Details: A total of 32 patients consented to participate, 5 patients failed screening and 2 did not receive any study drug. A total of 25 patients received at least one dose of study drug.
Groups:
- Cantrixil 0.24 mg/kg: Participants received Cantrixil 0.24 mg/kg administered as a single intraperitoneal dose once a week for up to 24 weeks (8 x 3-week cycles).
  In cycles 1-2 (6 weeks) they received Cantrixil only and in cycles 3-8 (18 weeks) they received Cantrixil in combination with a systemic chemotherapy.
- Cantrixil 0.6 mk/kg: Participants received Cantrixil 0.6 mg/kg administered as a single intraperitoneal dose once a week for up to 24 weeks (8 x 3-week cycles).
  In cycles 1-2 (6 weeks) they received Cantrixil only and in cycles 3-8 (18 weeks) they received Cantrixil in combination with a systemic chemotherapy.
- Cantrixil 1.25 mg/kg: Participants received Cantrixil 1.25 mg/kg administered as a single intraperitoneal dose once a week for up to 24 weeks (8 x 3-week cycles).
  In cycles 1-2 (6 weeks) they received Cantrixil only and in cycles 3-8 (18 weeks) they received Cantrixil in combination with a systemic chemotherapy.
- Cantrixil 2.5 mg/kg: Participants received Cantrixil 2.5 mg/kg administered as a single intraperitoneal dose once a week for up to 24 weeks (8 x 3-week cycles).
  In cycles 1-2 (6 weeks) they received Cantrixil only and in cycles 3-8 (18 weeks) they received Cantrixil in combination with a systemic chemotherapy.
- Cantrixil 5.0 mg/kg: Participants received Cantrixil 5.0 mg/kg administered as a single intraperitoneal dose once a week for up to 24 weeks (8 x 3-week cycles).
  In cycles 1-2 (6 weeks) they received Cantrixil only and in cycles 3-8 (18 weeks) they received Cantrixil in combination with a systemic chemotherapy.
- Cantrixil 10 mg/kg: Participants received Cantrixil 10 mg/kg administered as a single intraperitoneal dose once a week for up to 24 weeks (8 x 3-week cycles).
  In cycles 1-2 (6 weeks) they received Cantrixil only and in cycles 3-8 (18 weeks) they received Cantrixil in combination with a systemic chemotherapy.
- Cantrixil 20 mg/kg: Participants received Cantrixil 20 mg/kg administered as a single intraperitoneal dose once a week for up to 24 weeks (8 x 3-week cycles).
  In cycles 1-2 (6 weeks) they received Cantrixil only and in cycles 3-8 (18 weeks) they received Cantrixil in combination with a systemic chemotherapy.
Period: Part A: Dose Escalation Cohort
Arm/Group | Cantrixil 0.24 mg/kg | Cantrixil 0.6 mk/kg | Cantrixil 1.25 mg/kg | Cantrixil 2.5 mg/kg | Cantrixil 5.0 mg/kg | Cantrixil 10 mg/kg | Cantrixil 20 mg/kg
Started | 2 | 1 | 1 | 1 | 3 | 2 | 1
Completed (Completed 8 cycles of Cantrixil therapy) | 1 | 0 | 0 | 1 | 2 | 0 | 0
Not Completed | 1 | 1 | 1 | 0 | 1 | 2 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Progressive disease | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Part B: Expansion Cohort (5 mg/kg)
Arm/Group | Cantrixil 0.24 mg/kg | Cantrixil 0.6 mk/kg | Cantrixil 1.25 mg/kg | Cantrixil 2.5 mg/kg | Cantrixil 5.0 mg/kg | Cantrixil 10 mg/kg | Cantrixil 20 mg/kg
Started | 0 | 0 | 0 | 0 | 14 | 0 | 0
Completed (Completed 8 cycles of Cantrixil therapy) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 12 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Death due to progressive disease | 0 | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cantrixil 0.6 mg/kg: Participants received Cantrixil 0.6 mg/kg administered as a single intraperitoneal dose once a week for up to 24 weeks (8 x 3-week cycles).
  In cycles 1-2 (6 weeks) they received Cantrixil only and in cycles 3-8 (18 weeks) they received Cantrixil in combination with a systemic chemotherapy.
- Cantrixil 5 mg/kg: Participants received Cantrixil 5 mg/kg administered as a single intraperitoneal dose once a week for up to 24 weeks (8 x 3-week cycles).
  In cycles 1-2 (6 weeks) they received Cantrixil only and in cycles 3-8 (18 weeks) they received Cantrixil in combination with a systemic chemotherapy.
- Total: Total of all reporting groups
Arm/Group | Cantrixil 0.24 mg/kg | Cantrixil 0.6 mg/kg | Cantrixil 1.25 mg/kg | Cantrixil 2.5 mg/kg | Cantrixil 5 mg/kg | Cantrixil 10 mg/kg | Cantrixil 20 mg/kg | Total
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 17 | 2 | 1 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (18.38) | 70.0 (0) | 66.0 (0) | 66.0 (1) | 63.2 (8.63) | 65.0 (9.90) | 46.0 (0) | 62.5 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 1 | 17 | 2 | 1 | 25
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 4
  Not Hispanic or Latino | 2 | 1 | 1 | 1 | 13 | 2 | 1 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 1 | 1 | 16 | 2 | 1 | 23
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 0 | 0 | 0 | 0 | 10 | 1 | 1 | 12
  Australia | 2 | 1 | 1 | 1 | 7 | 1 | 0 | 13
Screening BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m2] | 25.29 (8.27) | 21.30 (0) | 25.50 (0) | 24.40 (0) | 27.98 (5.76) | 33.23 (7.14) | 38.2 (0) | 28.14 (6.061)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). Grade range 0-5; where 0 is best (no restrictions) and 5 is worst (dead)
  Participants
    0 (Fully active, able to carry on all pre-disease performance without restriction) | 2 | 1 | 0 | 1 | 6 | 2 | 0 | 12
    1 (Restricted in physically strenuous activity but ambulatory and able to carry out work activities) | 0 | 0 | 1 | 0 | 11 | 0 | 1 | 13
Tumor Stage at diagnosis [Count of Participants; unit: Participants] — Ovarian cancer stages range from stage I (1) through IV (4). Stages 1-2 mean it is early ovarian cancer.
  Stages 3-4 mean the cancer is advanced. The four stages of ovarian cancer may be divided into sub-stages, A, B, C, which indicate increasing amounts of tumour. The lower the number, the less the cancer has spread.
  Participants
    IC | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
    IIB | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
    IIIA | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    IIIB | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
    IIIC | 1 | 1 | 1 | 1 | 8 | 1 | 1 | 14
    IVA | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 5
    Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Tumor Stage at Study Entry [Count of Participants; unit: Participants] — Ovarian cancer stages range from stage I (1) through IV (4). Stages 1-2 mean it is early ovarian cancer. Stages 3-4 mean the cancer is advanced. The four stages of ovarian cancer may be divided into sub-stages, A, B, C, which indicate increasing amounts of tumour. The lower the number, the less the cancer has spread.
  Participants
    IIIA | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    IIIB | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
    IIIC | 0 | 1 | 0 | 0 | 4 | 1 | 1 | 7
    IVA | 2 | 0 | 0 | 0 | 7 | 0 | 0 | 9
    IVB | 0 | 0 | 1 | 0 | 4 | 1 | 0 | 6
Tumour Type [Count of Participants; unit: Participants]
  Ovarian Cancer | 2 | 1 | 1 | 1 | 11 | 1 | 1 | 18
  Fallopian Tube Cancer | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3
  Peritoneal Cancer | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 4
Histological Sub-Type [Count of Participants; unit: Participants]
  Serous Carcinoma | 2 | 0 | 0 | 1 | 11 | 2 | 1 | 17
  Endometrioid Carcinoma | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Clear Cell Carcinoma | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Other | 0 | 1 | 1 | 0 | 4 | 0 | 0 | 6
Grade [Count of Participants; unit: Participants] — The Grade describes how the cancer cells look compared to normal cells under a microscope. The grade suggests how quickly the cancer may grow, high grade cells suggested that the cancers cells will grow faster.
  Participants
    Low grade | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    High grade | 2 | 1 | 1 | 1 | 17 | 2 | 1 | 25
Prior lines of therapy [Mean (Standard Deviation); unit: Number of lines of previous therapy] — All patients had previous lines of anticancer therapies and previous lines of platinum therapy. For counting the number of previous lines of chemotherapy, the distinct number of chemotherapy regimens given in the Adjuvant, Neoadjuvant and Metastatic setting are considered.
  Number of lines of previous therapy | 2.5 (0.71) | 5.0 (0) | 2.0 (0) | 2.0 (0) | 4.0 (2.78) | 4.0 (2.83) | 2.0 (0) | 3.7 (2.48)
Prior bevacizumab [Count of Participants; unit: Participants] | 2 | 1 | 0 | 0 | 9 | 0 | 1 | 13
Patient Sensitivity to Platinum [Count of Participants; unit: Participants]
  Platinum-Sensitive | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 5
  Platinum-Resistant | 1 | 0 | 1 | 1 | 11 | 2 | 1 | 17
  Platinum-Refractory | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 3
Duration of Disease Diagnosis (months) [Mean (Standard Deviation); unit: months] | 49.15 (31.75) | 61.60 (0) | 17.20 (0) | 37.80 (0) | 62.59 (56.33) | 46.60 (8.63) | 34.70 (0.) | 56.27 (47.950)

OUTCOME MEASURES:

1. Primary Outcome: Determination of the Maximum Tolerated Dose (MTD)
Description: Determination of the MTD: At each dose level, the number and proportion of patients in the MTD population who experience a dose-limiting toxicity (DLT) during the DLT evaluation period (Cycle 1/Part A) of Cantrixil using standard safety monitoring assessments when administered as a monotherapy. The MDT was the dose level below the cohort in which 1 or more patients had experienced a DLT.
Time Frame: During Cycle 1 (21 days)
Population: The MTD population included all patients who experienced DLTs in Cycle 1/Part A, and those who received all 3 weekly doses of study treatment in Cycle 1/Part A. The safety data regarding the Cycle 1/Part A were used to determine MTD from this analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cantrixil 0.24 mg/kg | Cantrixil 0.6 mg/kg | Cantrixil 1.25 mg/kg | Cantrixil 2.5 mg/kg | Cantrixil 5 mg/kg | Cantrixil 10 mg/kg | Cantrixil 20 mg/kg
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 3 | 2 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0

2. Primary Outcome: Pharmacokinetic Profile
Description: Mean plasma concentration
Time Frame: Cycle 1, Day 1 (Monotherapy)
Population: All enrolled patients who received at least 1 dose of study treatment and who had undergone at least 1 PK assessment.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cantrixil 0.24 mg/kg | Cantrixil 0.6 mg/kg | Cantrixil 1.25 mg/kg | Cantrixil 2.5 mg/kg | Cantrixil 5 mg/kg | Cantrixil 10 mg/kg | Cantrixil 20 mg/kg
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 17 | 2 | 1
ng/ml
  Time (h): 0.00: number analyzed (Participants) | 2 | 1 | 1 | 1 | 15 | 1 | 1
  Time (h): 0.00 | 0.00 (0.00) | 0.00 | 0.00 | 0.00 | 0.00 (0.00) | 0.00 | 0.00
  Time (h): 0.083: number analyzed (Participants) | 2 | 1 | 1 | 1 | 16 | 2 | 1
  Time (h): 0.083 | 4.21 (5.95) | 43.8 | 52.2 | 73.9 | 227 (199) | 479 (304) | 5350
  Time (h): 0.5: number analyzed (Participants) | 2 | 1 | 1 | 1 | 16 | 1 | 1
  Time (h): 0.5 | 7.84 (1.68) | 62.4 | 84.9 | 202 | 279 (173) | 1220 | 6100
  Time (h): 1.00: number analyzed (Participants) | 2 | 1 | 0 | 1 | 16 | 2 | 1
  Time (h): 1.00 | 10.9 (3.13) | 53.8 |  | 217 | 262 (149) | 1150 (191) | 3830
  Time (h): 2.00: number analyzed (Participants) | 2 | 1 | 1 | 1 | 16 | 2 | 1
  Time (h): 2.00 | 13.1 (7.51) | 41.2 | 54.6 | 227 | 256 (161) | 1210 (205) | 3200
  Time (h): 4.00: number analyzed (Participants) | 2 | 1 | 0 | 1 | 16 | 2 | 1
  Time (h): 4.00 | 14.0 (5.86) | 24.8 |  | 187 | 207 (114) | 1080 (511) | 2400
  Time (h): 6.00: number analyzed (Participants) | 1 | 1 | 1 | 1 | 16 | 2 | 1
  Time (h): 6.00 | 15.0 | 13.2 | 41.2 | 162 | 170 (107) | 1030 (489) | 1040
  Time (h): 24.00: number analyzed (Participants) | 1 | 1 | 1 | 1 | 10 | 2 | 1
  Time (h): 24.00 | 0.971 | 0.0535 | 2.28 | 6.08 | 24.2 (17.1) | 20.7 (17.5) | 65.6

3. Primary Outcome: Pharmacokinetic Profile
Description: Mean plasma concentration
Time Frame: Cycle 3, Day 1 (Cantrixil plus chemotherapy)
Population: All enrolled patients who received at least 1 dose of study treatment and who had undergone at least 1 PK assessment.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cantrixil 0.24 mg/kg | Cantrixil 0.6 mg/kg | Cantrixil 1.25 mg/kg | Cantrixil 2.5 mg/kg | Cantrixil 5 mg/kg | Cantrixil 10 mg/kg | Cantrixil 20 mg/kg
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 17 | 2 | 1
ng/ml
  Time (h): 0.00: number analyzed (Participants) | 1 | 1 | 0 | 1 | 7 | 0 | 0
  Time (h): 0.00 | 0.00 | 0.00 |  | 0.00 | 0.258 (0.479) |  |
  Time (h): 0.083: number analyzed (Participants) | 1 | 1 | 0 | 1 | 6 | 0 | 0
  Time (h): 0.083 | 12.0 | 37.5 |  | 201 | 242 (106) |  |
  Time (h): 0.5: number analyzed (Participants) | 1 | 1 | 0 | 1 | 6 | 0 | 0
  Time (h): 0.5 | 18.5 | 48.7 |  | 261 | 368 (236) |  |
  Time (h): 1.00: number analyzed (Participants) | 1 | 1 | 0 | 1 | 7 | 0 | 0
  Time (h): 1.00 | 19.6 | 53.2 |  | 298 | 327 (210) |  |
  Time (h): 2.00: number analyzed (Participants) | 1 | 1 | 0 | 1 | 6 | 0 | 0
  Time (h): 2.00 | 20.2 | 45.1 |  | 193 | 298 (91.1) |  |
  Time (h): 4.00: number analyzed (Participants) | 1 | 1 | 0 | 1 | 7 | 0 | 0
  Time (h): 4.00 | 21.5 | 32.2 |  | 129 | 210 (129) |  |
  Time (h): 6.00: number analyzed (Participants) | 1 | 1 | 0 | 1 | 7 | 0 | 0
  Time (h): 6.00 | 19.8 | 22.3 |  | 112 | 174 (130) |  |
  Time (h): 24.00: number analyzed (Participants) | 0 | 1 | 0 | 1 | 6 | 0 | 0
  Time (h): 24.00 |  | 0.093 |  | 1.11 | 11.4 (10.2) |  |

4. Primary Outcome: Pharmacokinetic Profile
Description: Mean plasma concentration
Time Frame: Cycle 3, Day 8 (Cantrixil plus chemotherapy)
Population: All enrolled patients who received at least 1 dose of study treatment and who had undergone at least 1 PK assessment.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cantrixil 0.24 mg/kg | Cantrixil 0.6 mg/kg | Cantrixil 1.25 mg/kg | Cantrixil 2.5 mg/kg | Cantrixil 5 mg/kg | Cantrixil 10 mg/kg | Cantrixil 20 mg/kg
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 17 | 2 | 1
ng/ml
  Time (h): 0.00: number analyzed (Participants) | 1 | 1 | 0 | 1 | 7 | 0 | 0
  Time (h): 0.00 | 0.00 | 0.00 |  | 0.00 | 0.347 (0.918) |  |
  Time (h): 0.083: number analyzed (Participants) | 1 | 1 | 0 | 1 | 6 | 0 | 0
  Time (h): 0.083 | 6.04 | 17.5 |  | 429 | 290 (171) |  |
  Time (h): 0.5: number analyzed (Participants) | 1 | 1 | 0 | 1 | 6 | 0 | 0
  Time (h): 0.5 | 15.5 | 87.9 |  | 328 | 430 (166) |  |
  Time (h): 1.00: number analyzed (Participants) | 1 | 1 | 0 | 1 | 7 | 0 | 0
  Time (h): 1.00 | 19.3 | 75.5 |  | 243 | 309 (191) |  |
  Time (h): 2.00: number analyzed (Participants) | 1 | 1 | 0 | 1 | 7 | 0 | 0
  Time (h): 2.00 | 18.9 | 59.7 |  | 197 | 259 (168) |  |
  Time (h): 4.00: number analyzed (Participants) | 1 | 1 | 0 | 1 | 7 | 0 | 0
  Time (h): 4.00 | 17.1 | 31.1 |  | 129 | 204 (139) |  |
  Time (h): 6.00: number analyzed (Participants) | 0 | 1 | 0 | 1 | 7 | 0 | 0
  Time (h): 6.00 |  | 24.0 |  | 104 | 163 (142) |  |
  Time (h): 24.00: number analyzed (Participants) | 0 | 1 | 0 | 1 | 7 | 0 | 0
  Time (h): 24.00 |  | 0.0582 |  | 2.48 | 13.0 (11.0) |  |

5. Secondary Outcome: Disease Response
Description: Tumors were assessment via radiological imaging (MRI or CT). The Gynecological Cancer Intergroup (GCIG) has published a detailed guidance on the criteria that could be used in clinical trial protocols to define progression and response in recurrent disease using Response Evaluation Criteria in Solid Tumours (RECIST 1.1) together with the serum marker CA-125 (Rustin et al., Int J Gynecol Cancer 2011;21: 419Y423 DOI: 10.1097/IGC.0b013e3182070f17). Validated algorithms were used to assess best overall response. These algorithms combine response criteria for CA125, target lesions (up to 5 measurable lesions, 2 per organ, as defined by RECIST 1.1), non-target lesions (include ascites and peritoneal thickening, which are not measurable by RECIST 1.1), and new lesions (Yes/No). Example: a best overall response of complete response (CR) required the following composite scoring: Target lesion, CR + Non-Target lesion, CR + New lesions, no + CA-125, Normal.
Time Frame: Baseline to End of Study (maximum 36 weeks)
Population: The Full Analysis Population (FAS) included all enrolled patients, from Part A and Part B, who received at least 1 dose of study treatment and from whom at least 1 post-baseline efficacy measurement was obtained. Of the 25 patients, 9 were excluded from efficacy analyses, these were from dose groups: 0.24 mg/kg [n=1], 5 mg/kg [n=7]), 20 mg/kg [n=1].
Measure: Count of Participants; unit: Participants
Arm/Group | Cantrixil 0.24 mg/kg | Cantrixil 0.6 mg/kg | Cantrixil 1.25 mg/kg | Cantrixil 2.5 mg/kg | Cantrixil 5 mg/kg | Cantrixil 10 mg/kg | Cantrixil 20 mg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 10 | 2 | 0
Participants
  Complete response | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Partial response | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Progressive disease | 0 | 1 | 1 | 0 | 4 | 1 | 0
  Stable disease | 1 | 0 | 0 | 0 | 5 | 0 | 0

6. Secondary Outcome: Progression Free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum or the longest diameter of target lesion; or any new lesions (measurable or non-measurable) and Gynecological Cancer Intergroup (GCIG) criteria progression based on serum CA 125, as an increase equal to or greater than 2 the the upper limit of normal documented on 2 occasions.
Time Frame: Baseline to End of Study (maximum 36 weeks)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Cantrixil 20 mg/kg: Participants received Cantrixil 0.24 mg/kg administered as a single intraperitoneal dose once a week for up to 24 weeks (8 x 3-week cycles). In cycles 1-2 (6 weeks) they received Cantrixil only and in cycles 3-8 (18 weeks) they received Cantrixil in combination with a systemic chemotherapy.
Arm/Group | Cantrixil 0.24 mg/kg | Cantrixil 0.6 mg/kg | Cantrixil 1.25 mg/kg | Cantrixil 2.5 mg/kg | Cantrixil 5 mg/kg | Cantrixil 10 mg/kg | Cantrixil 20 mg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 10 | 2 | 0
Months
  RECIST 1.1: number analyzed (Participants) | 1 | 1 | 1 | 0 | 10 | 2 | 0
  RECIST 1.1 | 5.52 [NA to NA] — The upper 95% confidence limit was not estimable due to insufficient number of participants with events | 1.18 [NA to NA] — The upper 95% confidence limit was not estimable due to insufficient number of participants with events | 1.02 [NA to NA] — The upper 95% confidence limit was not estimable due to insufficient number of participants with events |  | 3.06 [1.22 to NA] — The upper 95% confidence limit was not estimable due to insufficient number of participants with events | 1.38 [1.38 to NA] — The upper 95% confidence limit was not estimable due to insufficient number of participants with events |
  RECIST 1.1 and GCIG: number analyzed (Participants) | 1 | 1 | 1 | 0 | 10 | 2 | 0
  RECIST 1.1 and GCIG | 5.52 [NA to NA] — The upper 95% confidence limit was not estimable due to insufficient number of participants with events | 1.18 [NA to NA] — The upper 95% confidence limit was not estimable due to insufficient number of participants with events | 1.02 [NA to NA] — The upper 95% confidence limit was not estimable due to insufficient number of participants with events |  | 3.06 [1.22 to 7.92] | 1.38 [1.38 to NA] — The upper 95% confidence limit was not estimable due to insufficient number of participants with events |

7. Secondary Outcome: Paracentesis Events
Description: Number of patients who experienced one or more paracentesis events
Time Frame: Baseline to End of Study (maximum 36 weeks)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cantrixil 0.24 mg/kg | Cantrixil 0.6 mg/kg | Cantrixil 1.25 mg/kg | Cantrixil 2.5 mg/kg | Cantrixil 5 mg/kg | Cantrixil 10 mg/kg | Cantrixil 20 mg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 10 | 2 | 0
Participants | 0 | 0 | 0 | 0 | 4 | 0 | 0

8. Secondary Outcome: CA-125 Level
Description: Concentration of CA-125 in peripheral blood
Time Frame: Baseline and End of Therapy (maximum 36 weeks)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Cantrixil 0.24 mg/kg | Cantrixil 0.6 mg/kg | Cantrixil 1.25 mg/kg | Cantrixil 2.5 mg/kg | Cantrixil 5 mg/kg | Cantrixil 10 mg/kg | Cantrixil 20 mg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 10 | 2 | 0
U/mL
  Baseline | 28.00 | 130.00 | 5.00 | 41.00 | 487.76 (599.07) | 51.50 (60.1) |
  End of therapy | 42.00 | 94.00 | 7.00 | 23.00 | 1153.17 (1577.828) | 96.50 (108.187) |

9. Other Pre Specified Outcome: Clonogenicity of Circulating Epithelial Tumour Cells (CETC)
Description: Clonogenicity of CETCs in peripheral blood and malignant ascites (if present), assayed using the MAINTRAC® CETC Count method by Genostics or similar methodology.
Time Frame: Baseline, End of Monotherapy (up to 6 weeks), End of Combination Therapy (up to 24 weeks)
Population: Stem cell marker analysis was conducted only amongst patients enrolled into PART A of the study. Data were not available for all patients, missing data were not imputed.
Measure: Mean (Standard Deviation); unit: Number of spheroid cells
Arm/Group | Cantrixil 0.24 mg/kg | Cantrixil 0.6 mg/kg | Cantrixil 1.25 mg/kg | Cantrixil 2.5 mg/kg | Cantrixil 5 mg/kg | Cantrixil 10 mg/kg | Cantrixil 20 mg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 2 | 1
Number of spheroid cells
  Baseline: number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 2 | 0
  Baseline | 73.0 | 0.0 | 2650.0 | 0.0 | 333.3 (305.51) | 0.0 (0.00) |
  End of mono therapy: number analyzed (Participants) | 0 | 1 | 0 | 1 | 2 | 1 | 0
  End of mono therapy |  | 0.0 |  | 0.0 | 325.0 (388.91) | 50.0 |
  End of therapy: number analyzed (Participants) | 0 | 0 | 0 | 1 | 3 | 0 | 0
  End of therapy |  |  |  | 0.0 | 0.0 (0.00) |  |

10. Other Pre Specified Outcome: Enumeration of Circulating Epithelial Tumour Cells (CETC)
Description: Number of CETC in peripheral blood and malignant ascites (if present), assayed using the MAINTRAC® CETC Count method by Genostics or similar methodology.
Time Frame: Baseline, End of Monotherapy (up to 6 weeks), End of Combination Therapy (up to 24 weeks)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: cells/mL
Arm/Group | Cantrixil 0.24 mg/kg | Cantrixil 0.6 mg/kg | Cantrixil 1.25 mg/kg | Cantrixil 2.5 mg/kg | Cantrixil 5 mg/kg | Cantrixil 10 mg/kg | Cantrixil 20 mg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 2 | 1
cells/mL
  Baseline: number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 2 | 0
  Baseline | 550.0 | 0.0 (0.0) | 50.0 | 0.0 (0.0) | 116.7 (125.83) | 0.0 (0.0) |
  End of mono therapy: number analyzed (Participants) | 0 | 1 | 0 | 1 | 2 | 1 | 0
  End of mono therapy |  | 300.0 |  | 400.0 | 150.0 (70.71) | 2200.0 |
  End of therapy: number analyzed (Participants) | 1 | 0 | 0 | 1 | 3 | 0 | 0
  End of therapy | 150.0 |  |  | 0.0 | 233.3 (104.08) |  |

11. Other Pre Specified Outcome: Expression of Stem Cell Markers: Aldehyde Dehydrogenase (ALDH)
Description: Expression of stem cell markers ALDH in the isolated colonies will be measured using fluorescein isothiocyanate-labelled (FITC-labelled) or alternatively labelled antibodies and scanning fluorescent microscopy techniques.
Time Frame: Baseline, End of Monotherapy (up to 6 weeks)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Number of ALDH expressing cells
Arm/Group | Cantrixil 0.24 mg/kg | Cantrixil 0.6 mg/kg | Cantrixil 1.25 mg/kg | Cantrixil 2.5 mg/kg | Cantrixil 5 mg/kg | Cantrixil 10 mg/kg | Cantrixil 20 mg/kg
Number analyzed (Participants) | 1 | 0 | 1 | 0 | 2 | 0 | 0
Number of ALDH expressing cells
  Baseline: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 0 | 0
  Baseline | 100.0 |  | 2650.0 |  | 81.0 |  |
  End of mono therapy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 0
  End of mono therapy |  |  |  |  | 80.0 (28.28) |  |

12. Other Pre Specified Outcome: Expression of Stem Cell Markers: CD44 Cells
Description: Expression of stem cell markers CD44 in the isolated colonies will be measured using fluorescein isothiocyanate-labelled (FITC-labelled) or alternatively labelled antibodies and scanning fluorescent microscopy techniques.
Time Frame: Baseline, End of Monotherapy (up to 6 weeks)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage of CD44 cells
Arm/Group | Cantrixil 0.24 mg/kg | Cantrixil 0.6 mg/kg | Cantrixil 1.25 mg/kg | Cantrixil 2.5 mg/kg | Cantrixil 5 mg/kg | Cantrixil 10 mg/kg | Cantrixil 20 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 0
percentage of CD44 cells
  Baseline: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Baseline |  |  |  |  | 95.0 |  |
  End of mono therapy |  |  |  |  | 87.5 (17.68) |  |

ADVERSE EVENTS:
Time Frame: Patients were followed from study entry up to 3 months after discontinuing therapy or until death or consent withdrawal, whichever occurred first, up to a maximum of 36 weeks.
Description: Adverse events were classified according to the MedDRA, Version 20.0. Adverse events were categorised for severity according to the NCI CTCAE Version 4.03
Groups:
- Cantrixil 20 mg/kg: Participants received Cantrixil 2- mg/kg administered as a single intraperitoneal dose once a week for up to 24 weeks (8 x 3-week cycles).
  In cycles 1-2 (6 weeks) they received Cantrixil only and in cycles 3-8 (18 weeks) they received Cantrixil in combination with a systemic chemotherapy.
Arm/Group | Cantrixil 0.24 mg/kg | Cantrixil 0.6 mg/kg | Cantrixil 1.25 mg/kg | Cantrixil 2.5 mg/kg | Cantrixil 5 mg/kg | Cantrixil 10 mg/kg | Cantrixil 20 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/1 | 0/1 | 2/17 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/1 | 1/1 | 0/1 | 13/17 | 2/2 | 1/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1 | 1/1 | 0/1 | 13/17 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cantrixil 0.24 mg/kg (N=2) | Cantrixil 0.6 mg/kg (N=1) | Cantrixil 1.25 mg/kg (N=1) | Cantrixil 2.5 mg/kg (N=1) | Cantrixil 5 mg/kg (N=17) | Cantrixil 10 mg/kg (N=2) | Cantrixil 20 mg/kg (N=1)
abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cantrixil 0.24 mg/kg (N=2) | Cantrixil 0.6 mg/kg (N=1) | Cantrixil 1.25 mg/kg (N=1) | Cantrixil 2.5 mg/kg (N=1) | Cantrixil 5 mg/kg (N=17) | Cantrixil 10 mg/kg (N=2) | Cantrixil 20 mg/kg (N=1)
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 6 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 7 | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 2 | 1
Fatigue (General disorders) | 2 | 0 | 0 | 0 | 4 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0

LIMITATIONS AND CAVEATS:
Small numbers of subjects analysed limit the data available for exploratory endpoints (circulating epithelial tumour cells, expression of stem cell markers, CD44 and aldehyde dehydrogenase).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT02903771/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT02903771/SAP_001.pdf